CLINICAL TRIAL: NCT04192812
Title: THE EFFICACY OF PREOPERATIVE USAGE OF GONADOTROPINE-RELEASING HORMONE AGONIST IN PATIENTS UNDERGOING TOTAL LAPAROSCOPIC HYSTERECTOMY DUE TO UTERIN FIBROIDS
Brief Title: PREOPERATIVE GONADOTROPINE-RELEASING HORMONE AGONIST THERAPY BEFORE SURGERY FOR UTERİN FIBROIDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alkü Alanya Education and Research Hospital (Other)
Responsible Party: Principal Investigator, MERAL TUĞBA ÇİMŞİR, ASSOCIATE PROFESSOR, Alkü Alanya Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ALKU RESEARCH HOSPİTAL
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Uterine Fibroid; Gonadotropin-Releasing Hormone-Dependent Precocious Puberty
MeSH Terms: conditions — Leiomyoma; Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Intervention Model Description: PROSPECTİVE RANDOMİSED CONTROLLED TRİAL
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnRHa (Experimental): 3,75 MG LEUPROLIDE ACETATE FOR EVERY 4 WEEKS THROUGHOUT 3 MONTHS BEFORE SURGERY
  Interventions: Drug: PREOPERATİVE GnRHa THERAPY (LEUPROLIDE ACETATE) BEFORE SURGERY FOR UTERİN FIBROIDS
- no GnRHa (Placebo Comparator): NO TREATMENT
  Interventions: Drug: NO GnRHa

INTERVENTIONS:
Drug: PREOPERATİVE GnRHa THERAPY (LEUPROLIDE ACETATE) BEFORE SURGERY FOR UTERİN FIBROIDS — THE EFFICACY OF PREOPERATIVE USAGE OF GnRHa IN PATIENTS UNDERGOING TOTAL LAPAROSCOPIC HYSTERECTOMY DUE TO UTERIN FIBROIDS
  Arms: GnRHa
Drug: NO GnRHa — THE EFFICACY OF PREOPERATIVE USAGE OF GnRHa IN PATIENTS UNDERGOING TOTAL LAPAROSCOPIC HYSTERECTOMY DUE TO UTERIN FIBROIDS
  Arms: no GnRHa

SUMMARY:
Uterin fibroids are the most common operation indication for hysterectomy. Dyring laparoscopic hysterectomy the amount of bleeding is a great difficulty.There are a lot of clinical researchs to reduce the haemorrhage during open hysterectomy but not laparoscopic procedure. In ALKU ERH clinic, researchers decided to smaller the size of fibroid by using GnRH analogues before total laparoscopic hysterectomy to reduce the haemorrhage amount.

DETAILED DESCRIPTION:
After randomising patients to two groups, one of the group will be controle group and the other group will be working group and researchers decided to use 3,75 mg leuprolide acetate as GnRHa subcutanously in every four week, throughout 3 months before surgery to the working group, researchers will record intraoperative amount of bleeding by measuring the blood in suction scale, the duration of surgery, difference between preoperative haemoglobin levels and uterin weight. researchers will comparise all theese parameters ibn to two groups.

ELIGIBILITY:
Inclusion Criteria:

* MYOMA UTERI
* APPROPİATE FOR LAPAROSCOPY

Exclusion Criteria:

* MALİGNANCY

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
AMOUNT OF BLEEDİNG | 0 minute - 180 minute
  WHOLE AMOUNT OF BLEEDING DURING SURGERY
DURATION AF SURGERY | 0 MINUTE- 180 MINUTE
  TIME BETWEEN INITIAL AND END OF SURGERY

CONTACTS AND LOCATIONS:
Overall Officials: MERAL TUĞBA ÇİMŞİR, Principal Investigator — ALKU EDUCATİON AND RESEARCH HOSPITAL
Locations (1):
- Alku Alanya Education and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 5 YEARS